CLINICAL TRIAL: NCT01227148
Title: Influence of Tightly Glucose Control on Hyperglycemic Toxicity and Protein
Brief Title: Influence of Tightly Glucose Control on Hyperglycemic Toxicity and Protein Catabolism in Critically Ill Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Chien-Wei Hsu, Kaohsiung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS95-070
Record Dates: First submitted 2010-10-15; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2006-04

CONDITIONS: Critically Ill Patients
Keywords: critical care, glycemic control, insulin, nitrogen balance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tightly glucose conntrol (Experimental)
  Interventions: Other: Tightly glucose control
- Conventional glucose control (Active Comparator)
  Interventions: Other: Conventional glucose control

INTERVENTIONS:
Other: Tightly glucose control — A continuous insulin infusion (50 IU of Actrapid HM) in 49.5 ml of 0.9 percent sodium chloride with the use of a pump was started when blood glucose level exceeded 140 mg/dl to maintain a blood glucose level of between 120 and 140 mg per deciliter. The dose of insulin was adjusted according to whole-blood glucose levels, measured at one-four-hour interval in arterial blood or arterial catheter was not available. The insulin dose was adjusted by a neuro-fuzzy method
  Other Names: euglycemic control
  Arms: Tightly glucose conntrol
Other: Conventional glucose control — a continuous insulin infusion was delivered when the blood glucose level exceeded 200 mg/dl and insulin level was then adjusted to maintain a blood glucose level of between 180 and 200 mg per deciliter.
  Other Names: conventional insulin therapy
  Arms: Conventional glucose control

SUMMARY:
To compare the differences of urinary nitrogen excretion, nitrogen balance and clinical outcomes between tightly insulin therapy and conventional insulin therapy in the ICU.

DETAILED DESCRIPTION:
Critical illness is associated with increased circulating concentrations of proinflammatory cytokines, such as tumor necrosis factor (TNF-α), interleukin (IL)-1, and IL-6 which may be important mediators of insulin resistance and results in hyperglycemia. Altered glucose metabolism was caused by release of counter regulatory hormones such as glucagons; epinephrine and cortisol oppose the normal action of insulin, leading to an increase in skeletal muscle proteolysis. It did not know whether tightly glucose control had beneficial effect in urinary nitrogen excretion and nitrogen balance.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the adult ICU who had baseline blood glucose > 180 mg/dl
* expected to require treatment in the ICU on 3 or more consecutive days.

Exclusion Criteria:

* pregnant patients
* patients with chronic renal loss (Chronic renal loss was defined as persistent acute renal failure, complete loss of kidney function > 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
24-hour urinary urea nitrogen(UUN)excretion, nitrogen balance and serum albumin and prealbumin. | up to the 14th study day

SECONDARY OUTCOMES:
ICU day, ventilator day, hospital day, episodes of acute renal injury, bacteremia, blood transfusion, gastrointestinal (GI) bleeding, hypoglycemia, and hospital mortality rate. | up to ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Wei Hsu, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Hsu CW, Sun SF, Lin SL, Huang HH, Wong KF. Moderate glucose control results in less negative nitrogen balances in medical intensive care unit patients: a randomized, controlled study. Crit Care. 2012 Dec 12;16(2):R56. doi: 10.1186/cc11299. PMID 22480187